CLINICAL TRIAL: NCT05862168
Title: Neoadjuvant Tislelizumab Combined With Albumin-paclitaxel, Cisplatin, and Fluorouracil in Patients With Locally Advanced Oral Squamous Cell Carcinoma ：A Single-arm, Prospective，Phase II Study
Brief Title: Neoadjuvant Treatment of Tislelizumab Combined Chemotherapy for Locally Advanced Oral Squamous Cell Carcinoma ：A Single-arm, Prospective, Phase II Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weijia Fang, MD (Other)
Responsible Party: Sponsor-Investigator, Weijia Fang, MD, Oncology Department director, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neo-TIME
Record Dates: First submitted 2023-05-07; First posted 2023-05-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Oral Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — tislelizumab; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Tislelizumab; Drug: Albumin paclitaxel; Drug: Cisplatin; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: Tislelizumab — The participants will receive 3 cycles of Tislelizumab, with 21 days each. 200mg of Tislelizumab will be used intravenously on the first day of each cycle.
Drug: Albumin paclitaxel — The participants will receive 3 cycles of Albumin paclitaxel, with 21 days each. 200mg/m^2 of Albumin paclitaxel will be used intravenously on the first day of each cycle.
Drug: Cisplatin — The participants will receive 3 cycles of Cisplatin, with 21 days each. 20mg/m^2 of Cisplatin will be used intravenously on days 1 through 3 of each cycle.
Drug: 5-Fluorouracil — The participants will receive 3 cycles of 5-Fluorouracil, with 21 days each. 600mg/m^2/d of 5-Fluorouracil will be used as a 120-hour continuous intravenous infusion on days 1 through 5.

SUMMARY:
TPF is still recommended as the preferred induction chemotherapy regimen for nonsurgical treatment of patients with LA HNSCC. Based on the KEYNOTE-048 study, all major guidelines recommend PD-1 monotherapy or PD-1 combined with chemotherapy as the new first-line standard treatment for patients with advanced HNSCC. The immunotherapy in operable LA HNSCC was also explored as neoadjuvant therapy due to the excellent data in advanced HNSCC. These explorations have also achieved good results. Therefore, this study aims to explore the pathological remission rate, the long-term benefit and safety of Tislelizumab combined with albumin paclitaxel, cisplatin and fluorouracil for locally advanced oral squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent form
2. Histopathological diagnosis of oral squamous cell carcinoma
3. Age: 18-75 years old , Gender: male and female
4. Primary tumor with a clinical stage of III/IVb (T1-2N+M0或T3-4N0-3M0, AJCC2018)
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS): 0-1
6. No previous systematic therapy for OSCC (including chemotherapy, EGFR inhibitors, VEGFR inhibitors such as bevacizumab, immune checkpoint inhibition such as anti-PD-1 or PD-L1 antibodies, anti-ctLA-4 antibodies, etc.);
7. Patients must have at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
8. Adequte organ function based on laboratory test values obtained during the screening period：1）Blood routine: white blood cells (WBCs) >3.0× 109/L, ANC >1.5× 109/L, platelets >75× 109/L, hemoglobin >9 g/L, 2）Liver function: alanine amino transferase/aspartate amino transferase (ALAT/ASAT) <2.5 times the upper limit of normal and bilirubin <1.5 times the upper limit of normal，3）Renal function: Serum creatinine <1.5 times the upper limit of normal，4）Coagulation function: INR, PT, APTT<1.5 times the upper limit of normal，5）Left ventricular ejection fraction (LVEF) ≥ 50%
9. contraception

Exclusion Criteria:

1. Known history of malignancy, unless been cured and no recurrence for 5 years
2. Patients with a history of active bleeding, coagulopathy, or receiving coumarin anticoagulation therapy
3. Known history of radiation, chemotherapy, surgery and immunology-based treatment to head and neck
4. Active autoimmune disease requiring systemic treatment within 2 years prior to the first dose, or autoimmune disease that may recur or plan treatment as judged by the investigator.
5. Active or previous definite inflammatory bowel disease (e.g., Crohn 's disease or ulcerative colitis) disease.
6. Subjects with known active pulmonary tuberculosis (TB) and suspected active TB require clinical examination to rule out; known active syphilis infection.
7. Serious infections within 4 weeks prior to the first dose, including but not limited to comorbidities requiring hospitalization, sepsis, or serious pneumonia; active infections (excluding antiviral therapy for hepatitis B or C) that have received systemic anti-infective therapy within 2 weeks prior to the first dose.
8. Known human immunodeficiency virus (HIV) infection
9. Subjects with untreated active hepatitis B (HBsAg positive and HBV-DNA more than 1000 copies/ml [200 IU/ml] or above the lower limit of detection) and anti-hepatitis B virus treatment during study treatment are required for subjects with hepatitis B; subjects with active hepatitis C (HCV antibody positive and HCV-RNA level above the lower limit of detection).
10. History of pneumonitis/interstitial lung disease requiring systemic corticosteroids or current pneumonitis.
11. Known allergic reaction to any ingredients or excipients of the therapy
12. Participation in other clinical trials within 30 days before enrollment
13. Pregnant or lactating women
14. Known alle Other situations that the investigator considers unsuitable with respect to participating in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response | 6 months

SECONDARY OUTCOMES:
Major pathologic response | 6 months
Event-free survival | 2 years
Disease-free survival | 5 years
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- First affiliated hospital, School of Medicine, Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No